CLINICAL TRIAL: NCT00581594
Title: Traditional vs. Graft-augmented Posterior Colporrhaphy: A Randomized Prospective Study
Brief Title: Traditional vs. Graft-augmented Posterior Colporrhaphy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not meet recruitment, technology advancement.
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-4574
Record Dates: First submitted 2007-12-20; First posted 2007-12-27 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Pelvic Organ Prolapse; Posterior Vaginal Wall Defects
Keywords: Pelvic organ prolapse; Posterior wall defects; Graft-augmented repair; Posterior colporrhaphy
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Posterior repair with graft augmentation.
  Interventions: Procedure: Graft-augmented colporrhaphy
- 2 (Other): Posterior repair without graft augmentation.
  Interventions: Procedure: Traditional posterior colporrhaphy

INTERVENTIONS:
Procedure: Graft-augmented colporrhaphy — Patients will undergo randomized surgical procedure. Patients will be seen at 6 weeks for a pelvic exam and evaluation of the posterior wall. Points Ap and Bp will be recorded with values at 0.5cm intervals being on the posterior vaginal wall that is 3cm above the hymen. Point Bp is the most dependent portion of the posterior vaginal wall when the patient performs a Valsalva maneuver. Patients will be seen at 6 months for a pelvic exam evaluation of posterior wall support and completion of SF-36, PISQ and FISI. Patients will be given 60 minute Questionnaires on defecatory dysfunction, pelvic pain and/or symptoms of prolapse. Patients will be seen at 1 year and yearly intervals up to five years for a pelvic exam for evaluation of posterior wall support and the questionnaires.
  Other Names: Xenform® material
  Arms: 1
Procedure: Traditional posterior colporrhaphy — Patients will undergo randomized surgical procedure. Patients will be seen at 2 weeks for routine post-op care and evaluation of any post-op complications. Patients will be seen at 6 weeks for a pelvic exam and evaluation of the posterior wall. Points Ap and Bp will be recorded with values at 0.5cm intervals being on the posterior vaginal wall that is 3cm above the hymen. Point Bp is the most dependent portion of the posterior vaginal wall when the patient performs a Valsalva maneuver. Patients will be seen at 6 months, for a pelvic exam evaluation of posterior wall support and completion of SF-36, PISQ and FISI. Patients will be given 60 minute Questionnaires on defecatory dysfunction, pelvic pain and/or symptoms of prolapse. Patients will be seen at 1 year and yearly intervals up to five years to have a pelvic exam for evaluation of posterior wall support and the questionnaires.
  Arms: 2

SUMMARY:
Women who undergo posterior colporrhaphy with graft augmentation will have a lower recurrence of their posterior wall defect than women who undergo a traditional posterior colporrhaphy.

DETAILED DESCRIPTION:
The traditional approach to surgical repair of posterior wall defect is the posterior colporrhaphy. Although this technique has been successful in the anatomic correction of the defect, the functional outcomes have been disappointing. This fact suggests improvement in the functional and anatomic outcomes following a traditional posterior colporrhaphy. Consequently, the idea of incorporating graft material into the repair to augment the patient's own tissue has been examined. Placing a piece of graft material in between the vagina and rectum adds an extra layer of support and thus augments the strength of the repair. The purpose of this study is to evaluate the anatomic and functional outcomes of posterior compartment, graft-augmented traditional posterior colporrhaphy vs. traditional posterior colporrhaphy alone.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Posterior wall defect with point Ap or Bp at 0 or greater
* Desires surgical correction
* Willing to accept randomization to graft vs. no graft
* Competent to sign an informed consent
* Completed childbearing
* Non-pregnant

Exclusion Criteria:

* Current anal sphincter disruption with planned incontinent surgical repairs
* Poor surgical candidate
* History of rectal cancer or inflammatory bowel disease
* Current rectovaginal
* History of vaginal cancer
* History of vaginal/pelvic radiation
* Foreshortened vagina
* Previous adverse reaction to Xenform matrix graft material

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-01; Primary Completion 2008-10-11 (Actual); Study Completion 2008-10-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome of recurrence of stage II posterior wall defects will be measured using the pelvic organ prolapse quantification exam (POPQ). | 5 Years

SECONDARY OUTCOMES:
The secondary outcomes will be measuring the effects of the surgical repair on various aspects of life using a series of questionnaires: SF-36 as a measure of quality of life, PISQ to measure sexual function, and FISI to measure rectal function. | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Noblett, M.D., Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States